CLINICAL TRIAL: NCT05353816
Title: Corheart 6 Left Ventricular Assist System Prospective, Multicenter, Single-arm Clinical Evaluation Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COREMED_LVAS
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-08

CONDITIONS: End-stage Heart Failure
Keywords: End-stage Heart Failure; Ventricular Assist System; Mechanical Circulatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corheart 6 LVAS (Experimental): Corheart 6 Left Ventricular Assist System (Corheart 6 LVAS) to be used on patients with end-stage heart failure.
  Interventions: Device: Corheart 6 Left Ventricular Assist System

INTERVENTIONS:
Device: Corheart 6 Left Ventricular Assist System — Implantation of the Corheart 6 Left Ventricular Assist Device for mechanical circulatory support.

SUMMARY:
This study is to evaluate the safety and effectiveness of the Corheart 6 Left Ventricular Assist System (Corheart 6 LVAS) used for the treatment of end-stage heart failure.

DETAILED DESCRIPTION:
The Corheart 6 Left Ventricular Assist System (also called "the Corheart 6 LVAS", or "the Corheart 6") is developed and manufactured by Shenzhen Core Medical Technology Co., Ltd. It is indicated for providing short-term and long-term mechanical circulatory support for patients with end-stage heart failure. This prospective, multi-center, and single-arm trial evaluates the safety and effectiveness of the device in treating patients with end-stage heart failure. 50 patients from 12 investigational sites will be enrolled for Corheart 6 VAS implantation and followed for 3 months post-implantation. Following the initial 3-month follow-up, the study was extended to assess the primary endpoint of event-free survival at 24 months, with further follow-up to 5 years to evaluate long-term outcomes. The primary endpoint include the success rate of device implantation at 3 months and event-free survival at 24 months post-implantation. All adverse events will be adjudicated by an independent Clinical Events Committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years.
* (2) The patient or legal representative has signed the Informed Consent Form (ICF).
* (3) Body Surface Area (BSA) ≥ 1.0 m^2.
* (4) Females of childbearing age must agree to use adequate contraception.
* (5) Patients with NYHA Class IV heart failure symptoms who have failed to be reversed by previous standardized oral treatment with anti-heart failure drugs (ACEI, beta-blockers, and diuretics).
* (6) Left Ventricular Ejection Fraction (LVEF) ≤ 30%, and at least one of the following conditions occurs:
* a. Fail to be reversed by or be weaned from intra-aortic balloon pump (IABP), extracorporeal membrane oxygenator (ECMO), or other short-term mechanical circulatory support;
* b. Rely on continuous intravenous administration of one or more vasoactive or inotropic drugs;
* c. Meeting the diagnostic criteria of cardiogenic shock: blood pressure < 90/60mmHg, cardiac index < 2.0 L/min/m^2, and pulmonary capillary wedge pressure > 18mmHg.

Exclusion Criteria:

* (1) Etiology of HF due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy pericardial disease, amyloidosis, or restrictive cardiomyopathy.
* (2) Presence of an active, uncontrolled infection confirmed by a combination of clinical symptoms and laboratory tests.
* (3) Technical obstacles which pose an inordinately high surgical risk, in the judgment of the investigator.
* (4) Intolerance to anticoagulant or antiplatelet therapies or any other peri/postoperative therapy the investigator will require based on the patient's health status.
* (5) Patients require bi-ventricular assist device support.
* (6) Pregnancy.
* (7) Presence of moderate to severe aortic insufficiency or a history of the mechanical aortic valve that will not be converted to a bioprosthesis or oversewn at the time of implantation.
* (8) History of any organ transplantation.
* (9) Presence of uncorrected thrombocytopenia or severe coagulopathy, such as diffuse intravascular coagulation.
* (10) TBIL (total bilirubin) > 3.0 mg/dL, serum creatinine (SCr) > 3.0 mg/dL within 48 hours prior to LVAD implantation surgery or may require dialysis.
* (11) History of severe chronic obstructive pulmonary disease (COPD) or restrictive lung disease or a diagnosis of primary pulmonary hypertension.
* (12) Pulmonary embolism and pulmonary artery systolic blood pressure exceeding 60mmHg within 3 weeks prior to enrollment combined with at least one of the following 2 parameters demonstrating that pulmonary vascular resistance did not respond to drug therapy: Pulmonary vascular resistance greater than 8 wood units; The transpulmonary differential pressure exceeds 20mmHg.
* (13) Established and untreated abdominal or thoracic aortic aneurysm > 5cm in diameter.
* (14) Presence of severe peripheral vascular disease with resting pain or extremity ulceration.
* (15) Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and Left Ventricular Assist System management, or brain death from various causes.
* (16) Expect to live less than 1 year due to malignant tumor or other diseases.
* (17) Participation in any other clinical trials that may influence the results of this study.
* (18) Other circumstances that are unforeseen and determined by the researcher to be unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
The success rate of device implantation at 3 months. | Up to 3 months post-implantation.
  The success rate of device implantation at 3 months post-implantation.
  Device implantation success will be met when a patient is still alive on device support, free of disabling stroke (modified Rankin Scale (mRS) > 3), and does not have the device replaced or removed due to device deficiency at 3 months post-implantation.
  The modified Rankin Scale is a tool used to assess functional disability or dependence in daily activities following a stroke or other neurological condition. It ranges from 0 (No observed neurological symptoms) to 6 (dead). Higher scores indicate more severe functional impairment.
The event-free survival at 24 months post-implantation. | Up to 24 months post-implantation
  Survival at 24 months post-implantation free of disabling stroke (mRS >3) or reoperation for device replacement. Subjects who undergo heart transplantation or device explantation due to myocardial recovery are considered to have met the primary endpoint.

SECONDARY OUTCOMES:
Functional status as measured by the New York Heart Association (NYHA) Classification | Baseline, at hospital discharge (within 5 days), and at 3, 6, 12, 24 and 60 months post-implantation.
  The NYHA (New York Heart Association) Functional Classification is a tool used to assess the severity of heart failure symptoms. It categorizes patients into one of four classes based on their level of activity limitation and symptoms. Class I represents no limitation of physical activity, while Class IV indicates severe limitations even at rest.
Quality of Life as measured by the EuroQoL-5D-3L (EQ-5D-3L) questionnaire | Baseline, at hospital discharge (within 5 days), and at 3, 6, 12, 24 and 60 months post-implantation.
  The EQ-5D-3L assesses health-related quality of life across five dimensions with three severity levels each. The scores from the 5 dimensions are summed for the total score which ranges from 5 to 15 with higher scores indicating more problems and a worse quality of life.
Quality of Life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ-23). | Baseline, at hospital discharge (within 5 days), and at 3, 6, 12, 24 and 60 months post-implantation.
  The Kansas City Cardiomyopathy Questionnaire (KCCQ-3) evaluates heart failure patients' health status, including symptoms, physical limitations, social limitations, self-efficacy, and quality of life. Scores range from 0 to 100, with higher scores indicating better health-related quality of life.
Functional status as measured by the Six Minute Walk Test (6MWT) | Baseline, at hospital discharge (within 5 days), and at 3, 6, 12, 24 and 60 months post-implantation.
  The 6-Minute Walk Test (6MWT) assesses functional capacity and endurance by measuring the distance walked in six minutes. Results vary based on age, gender, and disease severity. Generally, greater distances indicate better functional capacity and endurance.
Stroke severity as assessed with the National Institutes of Health Stroke Scale (NIHSS) score. | From baseline to 60 months post-implantation.
  The National Institutes of Health Stroke Scale measures stroke-related neurological deficits across various domains. Scores range from 0 to 42, with higher scores indicating more severe neurological impairment. Lower scores correlate with better neurological function.
Stroke severity as assessed by the modified Rankin Scale (mRS) score | From baseline to 60 months post-implantation.
  The modified Rankin Scale is a tool used to assess functional disability or dependence in daily activities following a stroke or other neurological condition. It ranges from 0 (No observed neurological symptoms) to 6 (dead). Higher scores indicate more severe functional impairment.
Adverse Events | From baseline to 60 months post-implantation.
  Frequency and incidence of all anticipated adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (11):
- China (11):
  - Fuwai Hospital, Chinese Academy of Medical Sciences(CAMS), Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second XIANGYA Hospital Of Central South University, Changsha, Hunan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Xijing Hospital of Air Force Medical University, Xi’an, Shanxi
  - People's Hospital of Xinjiang Uygur Autonomous Region, Xinjiang, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided
At this moment the IPD is not yet available for access and will be updated when it is ready.

REFERENCES:
- [Derived] Wang X, Chen H, Du J, Zhou X, Zou L, Huang J, Chen L, Cheng Z, Dong N, Chen X, Liu J, Yang Y, Wang C, Yang Y, Shen Z, Wang H, Hu S. A novel magnetically levitated intrapericardial left ventricular assist system in advanced heart failure-2-year results from a prospective, multi-centre study. Eur J Cardiothorac Surg. 2026 Jan 9:ezag014. doi: 10.1093/ejcts/ezag014. Online ahead of print. PMID 41512307